CLINICAL TRIAL: NCT06069375
Title: A Phase 2, Open-Label, Fixed Dose Study to Evaluate the Use of Sodium Phenylbutyrate (ACER-001) in the Treatment of Pediatric and Adult Patients With MCAD Deficiency Caused by the Common ACADM c.985 A>G (K304E) Mutation
Brief Title: Study of Sodium Phenylbutyrate (ACER-001) for the Treatment of Patients With Medium Chain Acyl-CoA Dehydrogenase Deficiency (MCADD)
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has been temporarily stopped until another study is completed. Data from the other study may inform changes to this study.
Sponsor: Jerry Vockley, MD, PhD (Other)
Collaborators: Acer Therapeutics Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jerry Vockley, MD, PhD, Chief, Division of Genetic and Genomic Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY23060034
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Medium-chain Acyl-CoA Dehydrogenase Deficiency
Keywords: Medium Chain Acyl-CoA Dehydrogenase Deficiency
MeSH Terms: conditions — Medium chain acyl CoA dehydrogenase deficiency | interventions — 4-phenylbutyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 3.0 g/m2/day QD sodium phenylbutyrate (Experimental): Up to 8 subjects (4 - ages 10-15 years old and 4 - 16 years of age and older) will be randomized to take 3.0 g/m2/day in one daily dose
  Interventions: Drug: Sodium phenylbutyrate
- 3.0 g/m2/day BID sodium phenylbutyrate (Experimental): Up to 8 subjects (4 - ages 10-15 years old and 4 - 16 years of age and older) will be randomized to take 3.0 g/m2/day divided into two daily doses taken 12 hours apart
  Interventions: Drug: Sodium phenylbutyrate
- 4.0 g/m2/day BID sodium phenylbutyrate (Experimental): Up to 8 subjects (4 - ages 10-15 years old and 4 - 16 years of age and older) will be randomized to take 4.0 g/m2/day divided into two daily doses taken 12 hours apart
  Interventions: Drug: Sodium phenylbutyrate

INTERVENTIONS:
Drug: Sodium phenylbutyrate — Open-label design with doses of sodium phenylbutyrate up to 4.0 g/m2/day
  Other Names: Olpruva

SUMMARY:
This is a medical research study to test a medication in patients 10 years of age and older with a disease called medium-chain acyl-CoA dehydrogenase deficiency (MCADD) caused by the common ACADM c.985 A>G (K304E) mutation. The medication is sodium phenylbutyrate (ACER-001), which is currently FDA approved for the treatment of Urea Cyle Disorders. Previous research suggests that sodium phenylbutyrate may also be effective in the treatment MCADD. This study will investigate the safety and efficacy (how well it works) of sodium phenylbutyrate in patients with MCADD.

DETAILED DESCRIPTION:
Participation in the study will require two overnight admissions and one outpatient visit at the Clinical and Translational Research Center at the UPMC Children's Hospital of Pittsburgh (also called the PCTRC). The total length of the study is 7 weeks.

Subjects will have blood work and an intravenous access line (IV) placed for several blood draws during the overnight visits. Subjects will begin fasting during the admission, which means they may consume only non-caloric fluids (water, unsweetened black coffee or tea, or sugar-free beverages). Bloodwork will be collected during the fast. Following the completion of the fast, the subject will eat a meal and will receive the study drug, sodium phenylbutyrate. The total time of fasting will be up to 24 hours for patients 16 years of age and older and up to 18 hours for patients 10-15 years of age.

Dosing for this study will be assigned to one of three doses: 3.0 g/m2/day in one daily dose, 3.0 g/m2/day divided into two daily doses 12 hours apart, and 4.0 g/m2/day divided into two daily doses 12 hours apart.

Subjects will return after 4 weeks to undergo the overnight admission and 18/24-hour fasting procedures outlined above. After the Week 5 admission they will no longer take the sodium phenylbutyrate.

Subjects will return after 2 weeks for an outpatient visit to have some additional blood work done and to make sure they are not experiencing any adverse effects.

All study procedures will be done at no cost to the subjects.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of MCADD and molecular confirmation of at least one copy of the common c.985A>G mutation.
* ≥16 years of age for cohort 1 and ≥10-15 years of age for cohort 2.
* Able to perform and comply with study activities including overnight admission to the PCTRC, placement of an IV catheter, and all blood draws.
* Negative pregnancy test for all female subjects of childbearing age.
* Signed informed consent by the subject or parent/guardian of minors.
* All females of childbearing age and all sexually active males must agree to use an acceptable method of contraception throughout the study. Appropriate contraceptive methods include hormonal contraceptives (oral, injected, implanted, or transdermal), tubal ligation, intrauterine device, hysterectomy, vasectomy, or double barrier methods. Abstinence is an acceptable form of birth control, though appropriate contraception must be used if the subject becomes sexually active.

Exclusion Criteria:

* Use of any investigational drug within 30 days of Day 1.
* Active infection (viral or bacterial) or any other intercurrent condition as reported by the subject or noted on physical exam at screening.
* Any clinical or laboratory abnormality of Grade 3 or greater severity according to the CTCAE v5.0, or Grade 3 elevations in liver enzymes, defined as levels 5-20 times ULN in alanine aminotransferase (ALT/SGPT), aspartate aminotransferase (AST/SGOT), or gamma glutamyl transpeptidase (GGT) in a clinically stable subject.
* Any clinical or laboratory abnormality or medical condition that, at the discretion of the investigator, may put the subject at increased risk by participating in this study.
* Use of any medication known to significantly affect renal clearance (e.g., probenecid) or to increase protein catabolism (e.g., corticosteroids), or other medication known to increase ammonia levels (e.g., valproic acid or haloperidol), within the 48 hours prior to Day 1 and throughout the study.
* Subjects with renal insufficiency will be excluded from the study. Cutoff eGFR <60 mL/min/1.73m2 (GFR categories G3a-G5) will be used as measure of renal insufficiency.
* Use of sodium benzoate within one week of Day 1.
* Known hypersensitivity to PAA or PBA.
* Breastfeeding or lactating females.
* Subjects at risk of hypokalemia due to pre-existing diagnosis or on medications that can cause hypokalemia.
* Subjects with type 1 or type 2 diabetes, or who take medications as part of their routine care that can cause hypoglycemia

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment related adverse events as assessed by CTCAE v5.0 | 7 weeks

SECONDARY OUTCOMES:
Length of fast before hypoglycemia develops | 4 weeks
  Comparision of the length of time each subject can fast, comparing their baseline fast to the fast after they are on sodium phenylbutyrate for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerard L Vockley, MD, PhD, Principal Investigator — UPMC Children's Hospital of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No